CLINICAL TRIAL: NCT01150097
Title: Extension Study to the Multicenter, Open-label, Randomized, Controlled Study CRAD001H2304 to Evaluate the Long-term Efficacy and Safety of Concentration-controlled Everolimus in Liver Transplant Recipient
Brief Title: Extension Study to Evaluate the Long-term Efficacy and Safety of Everolimus in Liver Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001H2304E1; 2009-017311-15
Record Dates: First submitted 2010-04-23; First posted 2010-06-24 (Estimated); Results first posted 2014-05-30 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Liver Transplant Recipient
Keywords: Liver transplantation; Everolimus; Calcineurin inhibitors; Tacrolimus; Renal function; Progression of HCV related allograft fibrosis
MeSH Terms: interventions — Tacrolimus; Everolimus; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Everolimus + reduced tacrolimus (Experimental): Participants were maintained on whole blood trough levels of 3 - 8 ng/mL everolimus and 3 - 5 ng/mL tacrolimus.
  Interventions: Drug: Tacrolimus (reduced tacrolimus); Drug: Everolimus (reduced tacrolimus); Drug: Corticosteroids
- Tacrolimus elimination (Experimental): Participants were maintained on a whole blood trough level of 6 - 10 ng/mL everolimus.
  Interventions: Drug: Tacrolimus (tacrolimus elimination); Drug: Everolimus (tacrolimus elimination); Drug: Corticosteroids
- Tacrolimus control (Active Comparator): Participants were maintained on a whole blood trough level of 6 - 10 ng/mL tacrolimus.
  Interventions: Drug: Tacrolimus (tacrolimus control); Drug: Corticosteroids

INTERVENTIONS:
Drug: Tacrolimus (reduced tacrolimus) — After everolimus whole blood trough levels were confirmed to be in the target range of 3-8 ng/mL, tacrolimus tapering began, achieving a target tacrolimus whole blood trough level of 3-5 ng/mL by 3 weeks after randomization, a level which was maintained for the duration of the study.
  Other Names: FK-506,; fujimycin,; Prograf,; Advagraf,; Protopic
  Arms: Everolimus + reduced tacrolimus
Drug: Everolimus (reduced tacrolimus) — Everolimus was started within 24 hours of randomization at a dose of 1.0 mg twice a day (bid, 2 mg daily dose). The dose was adjusted to maintain everolimus trough blood levels between 3-8 ng/mL for the duration of the study.
  Other Names: RAD001,; Zortress,; Certican,; Afinitor
  Arms: Everolimus + reduced tacrolimus
Drug: Tacrolimus (tacrolimus elimination) — After everolimus whole blood trough levels were confirmed to be in the target range of 3-8 ng/mL, tacrolimus tapering began, achieving a target tacrolimus whole blood trough level of 3-5 ng/mL by 3 weeks after randomization. Tacrolimus elimination was started beginning at Month 4. Tacrolimus was tapered after everolimus whole blood trough levels were within the target range of 6-10 ng/mL. Tacrolimus was completely eliminated by the end of Month 4.
  Other Names: FK-506,; fujimycin,; Prograf,; Advagraf,; Protopic
  Arms: Tacrolimus elimination
Drug: Everolimus (tacrolimus elimination) — Everolimus was started within 24 hours of randomization at a dose of 1.0 mg twice a day (bid, 2 mg daily dose). The dose was adjusted to maintain everolimus trough blood levels between 3-8 ng/mL until Month 4; beginning with Month 4, the dose was adjusted to maintain everolimus trough blood levels between 6-10 ng/mL.
  Other Names: RAD001,; Zortress,; Certican,; Afinitor
  Arms: Tacrolimus elimination
Drug: Tacrolimus (tacrolimus control) — Tacrolimus trough levels were targeted to be maintained at 8-12 ng/mL until Month 4. At Month 4, tacrolimus whole blood trough levels were decreased to a target trough level of 6-10 ng/mL for the remainder of the study.
  Other Names: FK-506,; fujimycin,; Prograf,; Advagraf,; Protopic
  Arms: Tacrolimus control
Drug: Corticosteroids — For patients in all groups, corticosteroids were initiated at or prior to the time of transplantation according to local practice. Corticosteroids could be used for the duration of the study but could not be eliminated before Month 6. The corticosteroids were not specified in the protocol because they were adminsitered to the participants according to local practice as part of standard of care.

SUMMARY:
The reason for this extension is to evaluate the long-term safety and efficacy of two concentration-controlled everolimus regimen in de novo liver transplant recipients. The most important long-term safety assessments include evaluation of renal function, progression of HCV related allograft fibrosis, and other treatment related effects at Month 36 post-transplantation compared to extension baseline (Months 24 post-transplantation).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Ability and willingness to adhere to study regimen
* Completed core study with assigned regimen;

Exclusion Criteria:

Patients fulfilling any of the following criteria are not eligible for inclusion in this study:

* Severe hypercholesterolemia or hypertriglyceridemia.
* Low platelet count.
* Low white blood cell count.
* Positive test for human immunodeficiency virus (HIV).
* Systemic infection requiring active use of IV antibiotics.
* Patients in a critical care setting.
* Use of prohibited medication.
* Use of immunosuppressive agents not utilized in the protocol.
* Hypersensitivity to any of the study drugs or similar drugs.
* Pregnant or nursing (lactating) women
* Women of child-bearing potential not using a highly effective method of birth control.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2010-03-31 (Actual); Primary Completion 2013-05-03 (Actual); Study Completion 2013-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (53):
- United States (13):
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Lexington, Kentucky
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Newark, New Jersey
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Houston, Texas
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, San Martín, Buenos Aires
- Australia (3):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Heidelberg, Victoria
- Belgium (3):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Brazil (2):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
- Colombia (2):
  - Novartis Investigative Site, Cali, Valle del Cauca Department
  - Novartis Investigative Site, Bogotá
- Novartis Investigative Site, Prague, Czech Republic, Czechia
- France (6):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Villejuif
- Germany (7):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
- Novartis Investigative Site, Dublin, Ireland
- Italy (5):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
- Novartis Investigative Site, Rotterdam, Netherlands
- Novartis Investigative Site, Moscow, Russia
- Spain (4):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barakaldo, Vizcaya
- Novartis Investigative Site, Stockholm, Sweden
- Novartis Investigative Site, Edinburgh, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two hundred eight four participants were eligible and enrolled into the extension. However, 2 participants withdrew from the extension prior to receiving treatment. Therefore, a total of 282 participants were accounted for in the extension.
Pre-assignment Details: Participants in the tacrolimus control group were studied for 12 months (from months 24 to 36 post transplant). Participants in the tacrolimus elimination and everolimus + reduced tacrolimus groups were studied for a minimum of 12 months up to 24 months (from months 24 to 48 months post transplant) depending on the participant's study start.
Period: Months 24 to 36 Post-transplantation
Arm/Group | Everolimus + Reduced Tacrolimus | Tacrolimus Elimination | Tacrolimus Control
Started | 106 | 51 | 125
Completed | 96 | 49 | 117
Not Completed | 10 | 2 | 8
Not completed — Death | 2 | 0 | 0
Not completed — Administrative problems | 5 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 3
Not completed — Withdrawal by Subject | 3 | 0 | 3
Period: Months 24 to 48 Post-transplantation
Arm/Group | Everolimus + Reduced Tacrolimus | Tacrolimus Elimination | Tacrolimus Control
Started | 106 | 51 | 0
Completed | 95 | 47 | 0
Not Completed | 11 | 4 | 0
Not completed — Administrative problems | 5 | 4 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Not completed — Death | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus + Reduced Tacrolimus | Tacrolimus Elimination | Tacrolimus Control | Total
Number analyzed (Participants) | 106 | 51 | 125 | 282
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (9.57) | 54.9 (10.07) | 55.2 (8.10) | 54.5 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 18 | 38 | 85
  Male | 77 | 33 | 87 | 197

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Composite Efficacy Failure Defined as Treated Biopsy Proven Acute Rejection (tBPAR ), Graft Loss or Death
Description: The number of participants who experienced composite efficacy failure was analyzed. Composite efficacy failure was defined as treated biopsy proven acute rejection (tBPAR), graft loss, or death. A BPAR was defined as an acute rejection confirmed by biopsy with a Rejection Activity Index (RAI) score ≥ 3. tBPAR was defined as a BPAR which was treated with anti-rejection therapy. The RAI is used to score liver biopsies with acute rejection and is composed of 3 categories (portal inflammation, bile duct inflammation damage, and venous endothelial inflammation) each scored on a scale of 0 (absent) to 3 (severe) by a trained pathologist. The total RAI score = the sum of the scores of the 3 categories and ranges from 0 to 9, with a higher score indicating greater rejection. The graft was presumed to be lost on the day the patient was newly listed for a liver graft, received a graft re-transplant, or died.
Time Frame: from months 24 to 36
Population: All extension participants
Measure: Number; unit: Participants
Arm/Group | Everolimus + Reduced Tacrolimus | Tacrolimus Elimination | Tacrolimus Control
Number analyzed (Participants) | 106 | 51 | 125
Participants | 2 | 1 | 3

2. Primary Outcome: Incidence Rate of Composite Efficacy Failure Defined as Treated Biopsy Proven Acute Rejection (tBPAR ), Graft Loss or Death
Description: as for outcome 1
Time Frame: from months 36 to 48
Population: Participants from the everolimus + reduced tacrolimus group and the tacrolimus elimination group
Measure: Number; unit: Participants
Arm/Group | Everolimus + Reduced Tacrolimus | Tacrolimus Elimination
Number analyzed (Participants) | 106 | 51
Participants | 1 | 0

3. Primary Outcome: Incidence Rate of Composite Efficacy Failure Defined as Graft Loss or Death
Description: The number of participants who experienced graft loss or death was analyzed. The graft was presumed to be lost on the day the patient was newly listed for a liver graft, received a graft re-transplant, or died.
Time Frame: from months 24 to 36
Population: All extension participants
Measure: Number; unit: Participants
Arm/Group | Everolimus + Reduced Tacrolimus | Tacrolimus Elimination | Tacrolimus Control
Number analyzed (Participants) | 106 | 51 | 125
Participants | 2 | 0 | 1

4. Primary Outcome: Incidence Rate of Composite Efficacy Failure Defined as Graft Loss or Death
Description: as for outcome 3
Time Frame: from months 36 - 48
Population: Participants from the everolimus + reduced tacrolimus group and the tacrolimus elimination group
Measure: Number; unit: Participants
Arm/Group | Everolimus + Reduced Tacrolimus | Tacrolimus Elimination
Number analyzed (Participants) | 106 | 51
Participants | 0 | 0

5. Secondary Outcome: Incidence Rate of tBPAR
Description: The number of participants who had a tBPAR was analyzed. tBPAR was defined as a BPAR which was treated with anti-rejection therapy. The RAI is used to score liver biopsies with acute rejection and is composed of 3 categories (portal inflammation, bile duct inflammation damage, and venous endothelial inflammation) each scored on a scale of 0 (absent) to 3 (severe) by a trained pathologist. The total RAI score = the sum of the scores of the 3 categories and ranges from 0 to 9, with a higher score indicating greater rejection.
Time Frame: from months 24 - 36
Population: All extension participants
Measure: Number; unit: Participants
Arm/Group | Everolimus + Reduced Tacrolimus | Tacrolimus Elimination | Tacrolimus Control
Number analyzed (Participants) | 106 | 51 | 125
Participants | 0 | 1 | 2

6. Primary Outcome: Change in Renal Function
Description: Change in renal function was assessed by the estimated Glomerular Filtration Rate (eGFR) using the abbreviated (4 variables) Modification of Diet in Renal Disease (MDRD-4) formula which was developed by the MDRD Study Group and has been validated in patients with chronic kidney disease. The MDRD-4 formula used for the eGFR calculation is: eGFR (mL/min/1.73m^2) = 186.3*(C^-1.154)*(A^-0.203)*G*R, where C is the serum concentration of creatinine (mg/dL), A is age (years), G=0.742 when gender is female, otherwise G=1, R=1.21 when race is black, otherwise R=1.
Time Frame: from months 24 to 36
Population: The analysis population included extension participants who had both post-extension baseline and month 36 values only.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Everolimus + Reduced Tacrolimus | Tacrolimus Elimination | Tacrolimus Control
Number analyzed (Participants) | 100 | 50 | 115
mL/min/1.73m^2 | -0.9 (16.13) | 2.5 (12.40) | -3.3 (11.84)

ADVERSE EVENTS:
Groups:
- Reduced TAC, Month 36: Reduced TAC, Month 36
- TAC Elimination, Month 36: TAC Elimination, Month 36
- TAC Control, Month 36: TAC Control, Month 36
- Reduced RAD + TAC, Month 48: Reduced RAD + TAC, Month 48
- TAC Elimination, Month 48: TAC Elimination, Month 48
Arm/Group | Reduced TAC, Month 36 | TAC Elimination, Month 36 | TAC Control, Month 36 | Reduced RAD + TAC, Month 48 | TAC Elimination, Month 48
Serious Adverse Events (participants affected / at risk) | 32/106 | 16/51 | 28/125 | 34/106 | 24/51
Other Adverse Events (participants affected / at risk) | 38/106 | 29/51 | 43/125 | 43/106 | 36/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reduced TAC, Month 36 (N=106) | TAC Elimination, Month 36 (N=51) | TAC Control, Month 36 (N=125) | Reduced RAD + TAC, Month 48 (N=106) | TAC Elimination, Month 48 (N=51)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 2 | 4 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 1
Device occlusion (General disorders) | 1 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0 | 1
Impaired healing (General disorders) | 2 | 1 | 0 | 2 | 2
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 2 | 2 | 3 | 4
Sudden death (General disorders) | 1 | 0 | 0 | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Biliary ischaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 1 | 0 | 1 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0
Hepatic artery thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatic necrosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 2 | 1
Epstein-Barr viraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0 | 1 | 2 | 0
Haematoma infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Orchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 2 | 3 | 3 | 3
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 2 | 1 | 0 | 2 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 1 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Wound abscess (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Graft loss (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 2 | 4
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reduced TAC, Month 36 (N=106) | TAC Elimination, Month 36 (N=51) | TAC Control, Month 36 (N=125) | Reduced RAD + TAC, Month 48 (N=106) | TAC Elimination, Month 48 (N=51)
Anaemia (Blood and lymphatic system disorders) | 4 | 3 | 3 | 4 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 8 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 10 | 3 | 4 | 13 | 4
Nausea (Gastrointestinal disorders) | 3 | 1 | 9 | 5 | 2
Fatigue (General disorders) | 1 | 2 | 10 | 2 | 6
Oedema peripheral (General disorders) | 4 | 4 | 2 | 6 | 5
Hepatitis C (Infections and infestations) | 1 | 2 | 3 | 1 | 3
Influenza (Infections and infestations) | 2 | 3 | 0 | 2 | 3
Nasopharyngitis (Infections and infestations) | 5 | 5 | 4 | 6 | 5
Urinary tract infection (Infections and infestations) | 4 | 2 | 4 | 4 | 4
Incisional hernia (Injury, poisoning and procedural complications) | 2 | 6 | 2 | 2 | 7
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 | 4 | 3 | 7 | 5
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 2 | 5
Renal failure (Renal and urinary disorders) | 1 | 1 | 10 | 2 | 1
Hypertension (Vascular disorders) | 8 | 2 | 5 | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.